CLINICAL TRIAL: NCT03438071
Title: Impact of Daily Videoconference Updates in Neonatal Intensive Care Unit on Parental Stress of Preterm Infants : a Pilot Study
Brief Title: Impact of Videoconference Updates in Neonatal Intensive Care Unit on Parental Stress of Preterm Infants (VISIO-NEONAT)
Status: Completed | Type: Observational
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: VISIO-NEONAT
Record Dates: First submitted 2018-02-04; First posted 2018-02-19 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Preterm Infants; Parent-Child Relations; Parental Stress; Post Partum Depression; Neonatal Intensive Care Units; Videoconferencing
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group
- Videoconference group
  Interventions: Other: Videoconferencing

INTERVENTIONS:
Other: Videoconferencing — Daily videoconference updates using Skype between parents of preterm infants hospitalized in NICU and the nurse taking care of their child, lasting 5 to 10 minutes, to check with her for the daily news and then see their child through the camera.
  Groups: Videoconference group

SUMMARY:
The aim of the study is to test the effect of daily videoconference updates between parents of preterm newborns and health care providers which also offer them the possibility of seeing their child on the parental stress in a neonatal intensive care unit (NICU).

ELIGIBILITY:
Inclusion Criteria:

* Parents with a preterm child born between 24 weeks and 34 weeks and 6 days of gestational age, hospitalized in our NICU during recrutment period
* Which agreed participating to the study after having complete information about it and sign a consent.

Exclusion Criteria:

* Parents with a preterm child with another pathology than prematurity or with a lenght of stay in the NICU less than 7 days
* Parents refusing to participate to the study
* Parents not having videoconference equipment or internet access at home
* Parents not understanding or speaking good enough French.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 30 preterm infants and their parents (15 in each group)
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2018-02-21 (Actual); Primary Completion 2018-08-18 (Actual); Study Completion 2018-09-07 (Actual)

PRIMARY OUTCOMES:
Level of stress of the mothers | From date of inclusion until the date of discharge, assessed up to 1 month
  Mean score of the mothers of preterm infants hospitalized in NICU on the PSS-NICU (Parental Stressor Scale NICU), measured once a week during all the last of their child's hospitalization in the unit, in the 2 groups.

SECONDARY OUTCOMES:
Level of stress of the fathers | From date of inclusion until the date of discharge, assessed up to 1 month
  Mean score of the fathers of preterm infants hospitalized in NICU on the PSS-NICU, measured once a week during all the last of their child's hospitalization in the unit, in the 2 groups.
Parental stress evolution | From the date of inclusion until the date of discharge, assessed up to 1 month
  Evolution of the PSS-NICU score of both parents between the inclusion in the study and the last evaluation before their child's discharge of the NICU, in the 2 groups.
Post-partum depression rate of the mothers | Through study completion, an average of 2 months
  Score of the mothers of preterm infants hospitalized in NICU on the EPDS (Edinburgh Post-natal Depression Scale), measured at the inclusion, at discharge and a month later, in the 2 groups.
Quality of the relationship between the parents and their child | Through study completion, an average of 2 months
  Mean score of both parents of preterm infants hospitalized in NICU on the PBQ (Post-partum Bonding Questionnaire), measured once a week during all the last of their child's hospitalization in the unit and a month after his discharge, in the 2 groups.

CONTACTS AND LOCATIONS:
Overall Officials: Denis Oriot, Principal Investigator — Poitiers University Hospital
Locations (1):
- CHU DE Poitiers, Poitiers, France

IPD SHARING:
Plan to Share IPD: No